CLINICAL TRIAL: NCT04852328
Title: Non-Randomized Phase 2 Trial of Three Schedules of CUE-101 Administered Before Surgery or Definitive Chemoradiation Therapy in HLA-A*0201 Positive Patients With Locally Advanced, HPV16-Positive Oropharyngeal Squamous-Cell Carcinoma
Brief Title: Three Schedules of CUE-101 Administered Before Surgery or Definitive Chemoradiation Therapy in HLA-A*0201 Positive Patients With Locally Advanced, HPV16-Positive Oropharyngeal Squamous-Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cue Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202106015
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Schedule A: CUE-101 (Experimental): * In Schedule A, CUE-101 will be administered during the neoadjuvant phase as a single dose given 14 days prior to initiation of standard of care (SOC) therapy.
  * Standard of care therapy consists of surgery and postoperative adjuvant (cisplatin) and radiation therapy or cisplatin and radiation therapy (definitive-chemoradiation therapy)
  Interventions: Drug: CUE-101
- Schedule B: CUE-101 (Experimental): * In Schedule B, CUE-101 will be administered during the neoadjuvant phase as two doses: one dose given 14 days and one dose given 7 days prior to initiation of standard of care (SOC) therapy.
  * Standard of care therapy consists of surgery and postoperative adjuvant (cisplatin) and radiation therapy or cisplatin and radiation therapy (definitive-chemoradiation therapy)
  Interventions: Drug: CUE-101
- Schedule C: CUE-101 (Experimental): * In Schedule C, CUE-101 will be administered during the neoadjuvant phase as a single dose given 7 days prior to initiation of standard of care (SOC) therapy.
  * Standard of care therapy consists of surgery and postoperative adjuvant (cisplatin) and radiation therapy or cisplatin and radiation therapy (definitive-chemoradiation therapy)
  Interventions: Drug: CUE-101

INTERVENTIONS:
Drug: CUE-101 — CUE Biopharma will supply CUE-101, which will be provided free of charge to the patient.

SUMMARY:
This is a phase 2 trial to assess the safety and tolerability of three schedules of CUE-101 administered in the neoadjuvant phase before standard of care (SOC) therapy to treatment naïve, HLA-A*0201 positive patients with newly diagnosed, locally advanced HPV16+ oropharyngeal squamous-cell carcinoma (OPSCC). This is an exploratory trial of a limited sample size to confirm safety and to assess for pharmacodynamic signals of efficacy in each of three schedules of CUE-101. Safety assessments will be performed at baseline and after CUE-101 administration. To assess for efficacy, peripheral blood and tumor samples will be collected at baseline and after CUE-101 administration. Following CUE-101, patients will proceed with SOC therapy, as prescribed by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous-cell carcinoma of the oropharynx or of an upper (levels 2-3) neck mass without a known primary site, but is suspected to be oropharynx based on clinical factors.
* Stage I-III (AJCC 8th Edition) [except clinical stages T1N0 and T2N0, which are excluded from enrollment].
* A candidate for standard of care therapy (either surgery followed by adjuvant therapy OR def-CRT), based on treating physician decision.
* HLA-A*0201 genotype as determined by genomic testing on blood sample performed at a CLIA-certified clinical or central laboratory.
* Tumors must test positive for HPV16 by PCR (performed on tumor) or ISH (performed in tumor) and p16INK4A expression (>70% staining in tumor cells) by IHC performed at a CLIA-certified clinical or central laboratory.
* Have archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion of sufficient size and quality for eligibility determination.
* At least 18 years of age.
* ECOG performance status ≤ 1.
* Normal bone marrow and organ function as defined below:

  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1,500/mcl
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Total bilirubin ≤ 1.5 x IULN, except patients with Gilbert's syndrome, who may enroll if the conjugated bilirubin (total and direct) is within normal limits
  * Creatinine < 1.5 mg/dL, or calculated or measured creatinine clearance >30 mL/min by Cockcroft-Gault
  * Note: Screening laboratory tests may be repeated once within 7 days.
* The effects of CUE-101 on the developing human fetus are unknown. For this reason and because novel Fc Fusion Protein agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 30 days after completion of the study.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* History of prior allogeneic bone marrow, stem-cell or solid organ transplantation
* Distant metastases.
* Treatment with radiation therapy or systemic anti-cancer therapy prior to the initiation of study drug administration.
* Treatment with corticosteroids (>10 mg per day prednisone or equivalent) or other immune suppressive drugs within the 14 days prior to the initiation of study drug administration. Corticosteroids for topical, ophthalmic, inhaled, or nasal administration are allowed. Physiological replacement with hydrocortisone up to a maximum dose of 40 mg per day is allowed.
* History of clinically significant cardiovascular disease including:

  * Myocardial infarction or unstable angina within the 16 weeks prior to the initiation of study drug
  * Clinically significant cardiac arrhythmias
  * Uncontrolled hypertension: systolic blood pressure >180 mmHg, diastolic blood pressure >100 mmHg
  * Deep vein thrombosis, pulmonary embolism, stroke, or transient ischemic attack within the 16 weeks prior to the initiation of study drug
  * QTc prolongation > 480 msec
  * Congestive heart failure (New York Heart Association class III- IV)
  * Pericarditis/clinically significant pericardial effusion
  * Myocarditis
* Clinically significant pulmonary compromise (eg, requirement for supplemental oxygen).
* Clinically significant gastrointestinal (GI) disorders including history of:

  * GI perforation within 1 year prior to study drug administration;
  * GI bleeding within 3 months prior to the initiation of study drug;
  * Acute pancreatitis within 3 months prior to the initiation of study drug;
  * Diverticulitis that is clinically significant in the opinion of the investigator based on the extent or severity of known disease and/or the occurrence of clinically significant disease flares within 4 weeks prior to the initiation of study drug administration; and/or
  * Cirrhosis.
* Evidence of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study drug. Patients requiring any systemic antiviral, antifungal, or antibacterial therapy for active infection must have completed treatment no less than 1 week prior to the initiation of study drug.
* Known history of hepatitis B or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction. However, patients with treated hepatitis C in complete remission and off therapy for > 1 year are eligible.
* Second primary invasive malignancy that has not been in remission for greater than 2 years. Exceptions include: non-melanoma skin cancer; cervical carcinoma in situ; squamous intraepithelial lesion on Pap smear; localized prostate cancer (Gleason score < 6); resected melanoma in situ; or favourable prognosis (<10% relapse risk) thyroid cancer.
* Prior treatment of the head and neck region with radiation therapy.
* History of major surgery within 4 weeks prior to the initiation of study drug administration. A diagnostic needle or excisional biopsy is not considered major surgery.
* Any serious underlying medical condition that would impair the ability of the patient to receive or tolerate the planned treatment at the investigational site.
* Known hypersensitivity to recombinant proteins, polysorbate 80 or any excipient contained in the drug formulation for CUE-101.
* Vaccination with any live virus vaccine within 4 weeks prior to the initiation of study drug administration. Inactivated annual influenza vaccination is allowed. Vaccination for COVID-19 is allowed within one week prior to initiation of study drug administration.
* Active or recent history of uncontrolled alcohol or other substance abuse within 3 months prior to the initiation of study drug administration.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 72 hours of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-related adverse events | From start of treatment through 12 months after the completion of standard of care treatment (estimated to be 15 months)
Number of adverse events | From start of treatment through 12 months after the completion of standard of care treatment (estimated to be 15 months
Treatment-related delays in start of standard of care therapy | From start of treatment through start of standard of care therapy (estimated to be 2 weeks)
  -Defined as >7 days of treatment-related delay from the planned date of surgery or initiation of definitive-chemoradiation therapy.
Change in frequency of HPV16 E711-20-specific CD8+ T cells in peripheral blood samples | Through 12 month follow-up
  * Determined by IFN γ ELISpot for detection of HPV16 E711-20-specific T cells
  * Baseline, prior to each CUE-101 infusion, 24 hours post-end of each CUE-101 infusion, prior to standard of care therapy, at day 28 post CUE-101, 2 month follow-up, 4 month follow-up, 8 month follow-up and 12 month follow-up
Change in frequency of HPV16 E711-20 tetramer-positive cytotoxic T cell lymphocytes | Through 12 month follow-up
  * Determined by multiparameter flow cytometry
  * Baseline, prior to each CUE-101 infusion, 24 hours post-end of each CUE-101 infusion, prior to standard of care therapy, at day 28 post CUE-101, 2 month follow-up, 4 month follow-up, 8 month follow-up and 12 month follow-up
Change in frequency of HPV16 E711-20-specific CD8+ T cells in tumor samples | Baseline, day -2 or -1 before start of standard of care therapy
Activation markers of HPV16 E711-20 tetramer-positive cytotoxic T cell lymphocytes | Through 12 month follow-up
Proliferative status of HPV16 E711-20 tetramer-positive cytotoxic T cell lymphocytes | Through 12 month follow-up

SECONDARY OUTCOMES:
Pathological tumor response | At the time of surgery or biopsy (Day 1 - approximately 7-14 days after start of CUE-101 treatment)
  * Defined as rates of major and complete pathological response
  * A major pathologic response (mPR) will be defined as ≤ 10% residual viable tumor within the tumor sample collected after administration of CUE-101. A complete pathologic response (cPR) will be defined as no invasive cancer in the tumor sample collected. For surgical patients, the tumor sample will include the primary tumor specimen and all sampled regional lymph nodes at the time of resection. For def-chemoradiation therapy patients, the tumor sample will comprise the biopsy(s) submitted. Pathologic tumor response will be stratified based on if the patients underwent surgery or post-CUE-101 biopsy only.
Objective response rate (ORR) | Prior to surgery/definitive chemoradiation treatment (Day 1 - approximately 7-14 after start of CUE-101 treatment)
  * Proportion of patients with a complete response + partial response
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Change in area under the concentration-time curve (AUC) of serum PK parameters | Through 12 month follow-up
  -Prior to each CUE-101 infusion, end of each CUE-101 infusion, 1 hour post-end of each CUE-101 infusion, 5 hours post-end of each CUE-101 infusion, 24 hours post-end of each CUE-101 infusion, surgery day 1 or definitive chemoradiation day -2 or -1, 2 month follow-up, 4 month follow-up, 8 month follow-up and 12 month follow-up.
Change in Cmax of serum PK parameters | Through 12 month follow-up
  -Prior to each CUE-101 infusion, end of each CUE-101 infusion, 1 hour post-end of each CUE-101 infusion, 5 hours post-end of each CUE-101 infusion, 24 hours post-end of each CUE-101 infusion, surgery day 1 or definitive chemoradiation day -2 or -1, 2 month follow-up, 4 month follow-up, 8 month follow-up and 12 month follow-up.
Change in Terminal elimination half-life(t1/2) of serum PK parameters | Through 12 month follow-up
  -Prior to each CUE-101 infusion, end of each CUE-101 infusion, 1 hour post-end of each CUE-101 infusion, 5 hours post-end of each CUE-101 infusion, 24 hours post-end of each CUE-101 infusion, surgery day 1 or definitive chemoradiation day -2 or -1, 2 month follow-up, 4 month follow-up, 8 month follow-up and 12 month follow-up.
Number of participants who relapse | Through 12 month follow-up
Number of participants who die summarized by cause of death | Through 12 month follow-up
Progression-free survival (PFS) | Through 12 month follow-up
Overall survival (OS) | Through 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu